CLINICAL TRIAL: NCT00114426
Title: Effects of Nocturnal Noninvasive Mechanical Ventilation on the Health Status of Patients With COPD
Brief Title: Effects of NIMV on the Health Status of Chronic Obstructive Pulmonary Disease (COPD )Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCT-52684
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2005-08-17 (Estimated); Status verified 2005-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: randomized controlled trial; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

INTERVENTIONS:
Device: non-invasive mechanical ventilation

SUMMARY:
In this proposal, we will implement a randomized controlled trial to determine whether nocturnal NIMV applied for 3 months: 1) improves (disease-specific) health related quality of life (HRQL) of COPD patients compared to a control group of patients treated with sham NIMV therapy (primary outcome); 2) improves exercise tolerance and walking capacity of COPD patients; and 3) improves heart rate variability and decreases sympathetic tone in COPD.

DETAILED DESCRIPTION:
COPD is one of the fastest growing conditions in the world, affecting over 16 million people in the US and over 1 million in Canada and costing society over $23 billion per annum (in the US). Its prevalence has risen by 41% since 1982, and the age-adjusted death rate has increased by 17% between 1966 and 1982 (in contrast to the decline in the age-adjusted death rates from all other causes during the same time period). By 2020, COPD will become the third leading cause of death (currently 4th representing 5% of all deaths worldwide) and 5th leading cause of disability (currently 12th) worldwide. Ironically, despite the rapidly growing public health burden of COPD, it is the most underfunded disease among all major causes of mortality in North America. Despite some progress in the management of COPD over the past two decades, there is still a paucity of efficacious therapies that can effectively modify the natural course of this disease.

There is a growing interest in nocturnal non-invasive mechanical ventilation (NIMV) therapy for long-term COPD management for several reasons. It may restore inspiratory rate, which diminishes by 30% during rapid eye movement (REM) sleep, improve gas exchange, and rest chronically tired respiratory muscles in COPD. Indeed, several uncontrolled studies have provided some empirical evidence to support the use of nocturnal NIMV in COPD. However, there is a paucity of well-designed controlled trials evaluating this novel therapy particularly for COPD patients at a high-risk for morbidity and mortality.

In this proposal, we will implement a randomized controlled trial to determine whether nocturnal NIMV applied for 3 months: 1) improves (disease-specific) health related quality of life (HRQL) of COPD patients compared to a control group of patients treated with sham NIMV therapy (primary outcome); 2) improves exercise tolerance and walking capacity of COPD patients; 3) reduces the number of clinical relapses in COPD patients; 4) improves heart rate variability and decreases sympathetic tone in COPD; and 5) is a "cost-effective" therapy.

We will carefully select COPD patients ready for discharge from an acute care hospital and will be invited to participate in this trial. Participants will then undergo a "run-in" phase of 4 weeks during which their clinical status will be stabilized. Patients experiencing a clinical exacerbation during the "run-in" phase will be excluded from the study. After the "run-in" phase, patients will be randomly assigned to one of two groups: nocturnal NIMV therapy + standard medical therapy or "sham" + standard medical therapy. The Chronic Respiratory Questionnaire (CRQ) and the Health Utilities Index Mark 2/3 (HUI 2 and HUI 3) will be used to measure HRQL of study participants at baseline and then at 2, 4, 6, 8, 10 and 12 weeks. We will also measure the study participants' exacerbation rate during the study period. A six-minute walk test will be used to determine the walking capacity of the study participants. In addition, 2-D echocardiography and 24-hour ambulatory electrocardiographic monitoring will be used to determine the effect of nocturnal NIMV on cardiac performance over a 3 month period. Finally, we will perform a comprehensive economic analysis to determine the costs as well as the benefits associated with the nocturnal NIMV therapy.

We anticipate that this study will show that those treated with nocturnal NIMV therapy will have better HRQL at 3 months compared to those on sham therapy and this will be associated with improved walking capacity and decreased rates of exacerbation. We also anticipate that nocturnal NIMV therapy will improve heart rate variability and lower pulmonary arterial pressure (during daytime).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of COPD and meeting the American Thoracic Society's definition of COPD
* Age 55 years of age or older;
* A history of 10 pack-years or more of cigarette smoking;
* FEV1 to FVC ratio of less than 70% and a postbronchodilator FEV1 of less than 50% of predicted (at baseline and after the run-in);
* PaC02 of 45 mm Hg or greater measured at rest on room air (at baseline and after run-in)

Exclusion Criteria:

* Coexisting medical conditions that make survival for at least 6 months unlikely;
* Refusal to participate;
* Cognitive impairment which makes it impossible to obtain informed consent;
* Patient on a lung transplant list;
* Clinical history of left ventricular heart failure;
* Body mass index of 35 kg/m2 or greater;
* (Obstructive) apnea-hypopnea index (AHI) of > 15 on polysomnography;
* Evidence of Cheyne-Stokes respiration on polysomnography;
* Impaired left ventricular ejection (LVEF of < 40% as determined on 2-D echocardiography);
* Patients who require rehospitalization, or an emergency visit for COPD during the run-in phase

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Health Status

SECONDARY OUTCOMES:
Heart Rate Variability

CONTACTS AND LOCATIONS:
Overall Officials: Don D Sin, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada